## **Study Protocol:**

The protocol of this randomized controlled clinical survey study was approved by the Ethical Committee of the Faculty of Dentistry, ondokuz mayıs university, Turkey, and the study was conducted in accordance with the Declaration of Helsinki. Informed written consent was obtained from all subjects after the details of the clinical procedures were explained. Systematically healthy 750 individuals (subject) aged ≥18 years that referred to the Department of Periodontology, Faculty of Dentistry, ondokuz mayıs University between 2015 and 2017, either for dental treatment or only for dental check-up were included in our study.

## Participants and assessments.

Prior to dental examination the questionnaire form to detect oral hygiene habits and oral hygiene consciousness levels and the OHIP-14 form to evaluate impact of periodontal status on quality of life were applied to each participants. The socio-demograhic data was recorded for each participant as age, sex, marital status, education level, monthly income.

Periodontal disease status was determined according to clinical and radiographic criteria. In order to determine the periodontal status of the plaque index(PI), gingival index (GI), probing pocket depth (PPD) and clinical attachment level (CAL) were recorded. Study participants were distributed into three groups as periodontally healthy(H; n=250), gingivitis (G; n=250)and chronic periodontitis (CP; n=250). The relationship between periodontal status with quality of life and perception of how oral health influences the quality of life as well as percieved oral health and oral hygiene consciousness level were evaluted.

## Assesment of perceived oral health and oral hygiene consciousness level.

The oral hygiene habits, frequency of dental visits and the age of first dental visit among the groups were recorded. Perceived oral health was measured by askin a question as 'How do you describe the health of your teeth and gums?' The patient based explanation of the periodontal status and the conciousness level about the application of oral hygiene measures were detected by asking 'What is the dental plaque for you?, What does plaque for you?, What is dental caries for you?, What is the dental calculus for you?, What is the symptom of bleeding from brushing teeth?, What is the cause of tooth and gum disease?, how do we

prevent tooth and gum disease?, What is the most important time of brushing?' in the questionnaire form.

## Assessment of OHIP 14 Scale.

The validity and reliability of OHIP, consisting of 49 questions, was made by Slade and Spencer (Slade, 1997). The short form of OHIP was developed due to answering and scoring scales can take a long time and the validity and reliability of OHIP-14 is confirmed by Slade (Slade, 1997; Nuttall, 2001). The answers are scored according to the Likert scale. Responses to the items were recorded on a six-point scale: never=0, seldom=1, sometimes=2, fairly often=3, very often=4 and all time=5 (Slade 1997). The high scores revealed the adversely affected quality of life (Slade,1997; Başol at al., 2014). The participants were informed on how to complete the indexes. Cronbach's alpha value, which indicates the internal consistency of the scale, is 0.94. The reliability and validity of the Turkish version of the OHIP-14 scale was determined by Mumcu et al. (2006) report.